CLINICAL TRIAL: NCT02511561
Title: A 1-Month, Prospective, Multicenter, Open-Label Study of OTO-201 Given as a Single Administration for Treatment of Otitis Externa
Brief Title: OTO-201 for the Treatment of Otitis Externa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201-201506
Record Dates: First submitted 2015-07-28; First posted 2015-07-30 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Otitis Externa
Keywords: Otitis externa; Swimmer's ear; Ear infection
MeSH Terms: conditions — Otitis Externa; Otitis | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.1 mL OTO-201 (Experimental): Ciprofloxacin
  Interventions: Drug: OTO-201 (ciprofloxacin)
- 0.2 mL OTO-201 (Experimental): Ciprofloxacin
  Interventions: Drug: OTO-201 (ciprofloxacin)
- 0.4 mL OTO-201 (Experimental): Ciprofloxacin
  Interventions: Drug: OTO-201 (ciprofloxacin)

INTERVENTIONS:
Drug: OTO-201 (ciprofloxacin)

SUMMARY:
This is a 1-month, multicenter, open-label study in subjects with unilateral otitis externa. Eligible subjects will receive a single dose of 6 mg OTO-201 to the affected ear. The study is designed to characterize safety, procedural factors and clinical effect of OTO-201 administered in subjects with otitis externa.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject is a male or female aged 6 months to 80 years, inclusive
* Subject has a clinical diagnosis of unilateral otitis externa
* Subject or subject's caregiver is willing to comply with the protocol and attend all study visits

Exclusion Criteria includes, but is not limited to:

* Subject has tympanic membrane perforation
* Subject has a history of known immunodeficiency disease
* Subject has fungal otitis externa, based on clinical signs

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl LeBel, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Email Otonomy Central Contact for Trial Locations, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 mg OTO-201: 6 mg ciprofloxacin: single administration
- 12 mg OTO-201: 12 mg ciprofloxacin: single administration
- 24 mg OTO-201: 24 mg ciprofloxacin: single administration
Period: Overall Study
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201 | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (21.95) | 30.0 (20.12) | 43.0 (23.74) | 37.3 (22.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 12 | 35
  Male | 13 | 14 | 13 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 2 | 12
  Not Hispanic or Latino | 21 | 19 | 23 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 5 | 11
  White | 22 | 21 | 18 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Otoscopic Examination: Tympanic Membrane
Description: Number of subjects with a tympanic membrane that was rated as "Not able to Visualize" or "Abnormal" at Baseline that was rated as "Normal" at Day 29 (final study day)
Time Frame: Up to 1 month
Population: Safety analysis set: All subjects who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 25 | 25 | 25
Participants | 6 | 8 | 8

2. Primary Outcome: Otoscopic Examination: Middle Ear
Description: Number of subjects with a middle ear that was rated as "Not Able to Visualize" or "Abnormal" at Baseline that had a middle ear rated as "Normal" at Day 29 (final study visit)
Time Frame: Up to 1 month
Population: Safety analysis set: All subjects that received drug
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 25 | 25 | 25
Participants | 8 | 7 | 8

3. Primary Outcome: Feasibility of Administration
Description: Ease of administering OTO-201 to the external ear canal. Number of subjects that investigators rated ease of administration as either "easy" or "very easy".
Time Frame: Day1
Population: Safety analysis set: All subjects who receieved study drug
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 25 | 25 | 25
Participants | 24 | 25 | 25

4. Primary Outcome: Overall Adverse Events
Description: Number of Subjects with and without adverse events during the study from dosing up to 1 month after dosing
Time Frame: up to 1 month
Population: Safety analysis set: All subjects that received study drug
Measure: Count of Participants; unit: Participants
Groups:
- 12 mg OTO-201: 12 ciprofloxacin: single administration
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 25 | 25 | 25
Participants
  Number of subjects with at least 1 adverse event | 8 | 9 | 13
  Number of subjects with no adverse events | 17 | 16 | 12

5. Secondary Outcome: Number of Subjects Considered a Clinical Cure at Day 15 (Intent-to-treat Analysis Set)
Description: Clinical Signs (edema, erythema, otorrhea and otalgia) all had a score of 0 at Day 15. Each sign was graded as follows:
  None = 0 Mild = 1 Moderate = 2 Severe = 3
Time Frame: Day 15 (two weeks from dosing)
Population: Intent-to-treat analysis set: All subjects who were randomized and were used for assessments of clinical activity
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 25 | 25 | 25
Participants | 14 | 19 | 16

6. Secondary Outcome: Number of Subjects Considered a Clinical Cure at Day 15 (Per-protocol Analysis Set)
Description: as for outcome 5
Time Frame: Day 15 (2 weeks from dosing)
Population: Per-protocol Analysis Set defined as all subjects in the ITT analysis set who received study drug, completed Visit 4 (Day 15), and did not have a major protocol deviation.
Measure: Count of Participants; unit: Participants
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
Number analyzed (Participants) | 24 | 22 | 25
Participants | 13 | 19 | 15

ADVERSE EVENTS:
Time Frame: Adverse events were reported during dosing and up to 1 month following dosing.
Arm/Group | 6 mg OTO-201 | 12 mg OTO-201 | 24 mg OTO-201
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 5/25 | 10/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 6 mg OTO-201 (N=25) | 12 mg OTO-201 (N=25) | 24 mg OTO-201 (N=25)
Otitis externa (Infections and infestations) | 2 | 3 | 4
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 3
Hypacusis (Ear and labyrinth disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication subject to Sponsor consent.